CLINICAL TRIAL: NCT06698393
Title: Impact of Different Polyamide Suture Diameter on Clinical Outcomes in Periodontal Plastic Surgery: a Randomized Controlled Trial
Brief Title: Different Suture Diameters in Periodontal Plastic Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Michele Paolantonio, Full Professor, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16112024
Record Dates: First submitted 2024-11-18; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Clinical Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Suture 3.0 Group (Active Comparator): Coronally Advanced Flap Combined with a Connective Tissue Graft Harvested from the Palate for the Treatment of RT1 Gingival Recession. The flap was repositioned using a non-resorbable polyamide suture with a diameter of 3.0
  Interventions: Procedure: Suture 3.0 Group
- Suture 6.0 Group (Experimental): Coronally Advanced Flap Combined with a Connective Tissue Graft Harvested from the Palate for the Treatment of RT1 Gingival Recession. The flap was repositioned using a non-resorbable polyamide suture with a diameter of 6.0
  Interventions: Procedure: Suture 6.0 Group

INTERVENTIONS:
Procedure: Suture 3.0 Group — The extent of the depth of the recession will be reported on the anatomical papillae and, after adding 1 mm, 2 horizontal incisions of approximately 3 mm will be made at the base of the surgical papillae laterally to the recession.Two divergent releasing incisions will be made extending approximately 2-3 mm into the alveolar mucosa.The surgical papillae will be detached in partial thickness. A full thickness dissection will be performed from the bottom of the recession to expose approximately 3mm of the crest bone.A partial thickness dissection will be performed in the most apical portion of the flap until complete passivation of the flap is obtained.The harvesting of the epithelial-connective graft will be performed at the la. The de-epithelialised graft will be sutured at the level of the de-epithelialised anatomical papillae.The flap will be repositioned coronally suturing the anatomical papillae on the surgical ones, using a Non-Resorbable Polyamide Suture of 3.0 Diameter.
  Arms: Suture 3.0 Group
Procedure: Suture 6.0 Group — The extent of the depth of the recession will be reported on the anatomical papillae and, after adding 1 mm, 2 horizontal incisions of approximately 3 mm will be made at the base of the surgical papillae laterally to the recession.Two divergent releasing incisions will be made extending approximately 2-3 mm into the alveolar mucosa.The surgical papillae will be detached in partial thickness. A full thickness dissection will be performed from the bottom of the recession to expose approximately 3mm of the crest bone.A partial thickness dissection will be performed in the most apical portion of the flap until complete passivation of the flap is obtained.The harvesting of the epithelial-connective graft will be performed at the la. The de-epithelialised graft will be sutured at the level of the de-epithelialised anatomical papillae.The flap will be repositioned coronally suturing the anatomical papillae on the surgical ones, using a Non-Resorbable Polyamide Suture of 6.0 Diameter.
  Arms: Suture 6.0 Group

SUMMARY:
This randomized controlled clinical trial aims to compare the clinical outcomes of using non-resorbable polyamide sutures of different diameters (3.0 vs. 6.0) for securing an advanced coronary flap (CAF) and subepithelial connective tissue graft (SCTG) in the treatment of RT1 gingival recessions (as classified by Cairo et al.).

Forty patients presenting with at least one RT1 recession will be enrolled in the study. Twenty participants will undergo CAF + SCTG sutured with non-resorbable polyamide thread of 3.0 diameter, while the other 20 participants (control group) will receive the same procedure sutured with a 6.0 diameter thread. The primary outcome, complete root coverage (CRC), will be assessed six months after treatment.

Additional clinical parameters, including gingival recession (GR), clinical attachment level (CAL), pocket depth (PD), keratinized tissue width (KT), keratinized tissue thickness (GT), and Root Coverage Esthetic Score (RES), will be evaluated at baseline and at the six-month follow-up.

Patient-reported outcomes (PROs) will also be measured, including the degree of general discomfort (D) experienced, assessed on a Visual Analog Scale (VAS) from 0 to 10, as well as patient-reported aesthetic satisfaction (PRES) and overall treatment satisfaction (OTS), both quantified on a VAS scale from 0 to 10.

DETAILED DESCRIPTION:
The study will be a prospective, randomized, and controlled clinical trial designed to compare two polyamide sutures of different diameters (3.0 and 6.0) used to secure a CAF + SCTG. For each study patient, one RT1 recession will be included. Clinical parameters will be evaluated at baseline and six months after treatment.

Forty patients under care at the Periodontology Unit of the University of Chieti-Pescara, Italy, and presenting RT1 recessions, will be selected for inclusion.

All 40 patients will first undergo professional supragingival scaling using ultrasonic instruments. Patients will also receive motivational oral hygiene instructions to adopt proper, pressure-free brushing techniques and non-traumatic use of dental floss and/or interdental brushes. The use of a pressure-controlled electric toothbrush with an extra-soft head will be recommended, and detailed instructions for its use will be provided. Access to the surgical phase will only be permitted after the achievement of supragingival plaque control through these non-traumatic oral hygiene procedures.

A computer-generated, customized randomization table will be used to allocate experimental units into the two study groups.

Post-surgical care will include a regimen of 2 g/day of amoxicillin combined with clavulanic acid for six days and oral ketoprofen as needed for pain control. Sutures will be removed two weeks after surgery. Plaque control of the grafted area will be managed for three weeks post-surgery with a twice-daily rinse using a 0.12% chlorhexidine digluconate solution. Additionally, patients will apply a 1% chlorhexidine gel twice daily. Patients will undergo weekly professional supragingival cleaning and motivational reinforcement sessions for six weeks. Gentle cleaning with a soft toothbrush and interdental cleaning will be allowed starting two weeks after suture removal. All measurements will be performed by a single experienced operator. Complete root coverage (CRC) will be assumed as the main outcome at 6 months after treatment. Gingival recession (GR), clinical attachment level (CAL), pocket depth (PD), keratinized tissue width (KT,) thickness of keratinized tissue (GT), Root coverage esthetic score will be assessed at baseline and 6 months after treatment. PROMs will also be evaluated. The degree of general discomfort (D) experienced will be assessed on a VAS scale (0-10). Patient-reported aesthetic satisfaction (PRES) at T1 will also be quantified on a VAS scale (0-10). Overall treatment satisfaction (OTS) at T1 will be assessed by asking each patient if they would undergo surgery again (yes/no).

ELIGIBILITY:
Inclusion Criteria:

* systemic factors (no systemic diseases; no coagulation disorders; no medications affecting periodontal status in the previous 6 months; no pregnancy or lactation
* never smokers/former smokers >=10years
* a full-mouth plaque score (FMPS)and a full-mouth bleeding score (FMBS) lower than 15%
* no periodontal surgery on the experimental sites
* >= 20 teeth without mobility
* no presence of cervical carious lesions or periapical lesions at experimental sites
* at least one RT1 buccal gingival recession

Exclusion Criteria:

* systemic diseases
* coagulation disorders
* medications affecting periodontal status in the previous 6 months
* pregnancy or lactation
* Smokers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Complete root coverage | 6 months
  Percentage of experimental sites that achieved complete root surface coverage.

SECONDARY OUTCOMES:
Gingival Recession | 6 months
  Distance from cementoenamel junction and gingival margin
Gingival thickness | 6 months
  Gingival tissue thickness evaluated 2 mm apical to the recession
Keratinized tissue width | 6 months
  Distance between gingival margin and Mucogingival Junction
Clinical attachment level | 6 months
  Distance between cementoenamel junction(CEJ) and depth of the pocket
Pocket depth | 6 months
  Distance between gingival margin and bottom of the pocket
Discomfort | 4 weeks
  Evaluation of post-operative discomfort using Visual Analogue Scale (VAS).The scale is represented by a straight horizontal line of fixed length, generally 10 cm. Extremities are defined as extreme limits of the parameter to be measured, oriented from left (worst) to right (best).
Patient-Reported Esthetic Satisfaction | 6 months
  Patient-reported esthetic satisfaction (PRES) quantified on a VAS scale (0-10), will be recorded after observing simultaneously 2 standardized photographs showing the treated site +2 mesial and 2 distal teeth and the MGJ
Root Coverage Esthetic Score | 6 months
  This score evaluates five variables: level of the gingival margin, marginal tissue contour, soft tissue texture, mucogingival junction alignment, and gingival color.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Innovative Technologies in Medicine and Dentistry, Chieti, Italy